CLINICAL TRIAL: NCT02946801
Title: Antiplaque Effect of Essential Oils and 0.2% Chlorhexidine on an in Situ Model of Oral Biofilm Growth. A Randomized Clinical Trial
Brief Title: Antiplaque Effect of Essential Oils With and Without Alcochol on an in Situ Model of Oral Biofilm Growth
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Inmaculada Tomas, Senior Lecturer, University of Santiago de Compostela
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 395/2016
Record Dates: First submitted 2016-10-21; First posted 2016-10-27 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Biofilms; Oils, Essential; Periodontitis
Keywords: Biofilms; essential oils; alcohol; microscopy, confocal; mouthwashes
MeSH Terms: conditions — Periodontitis | interventions — Oils, Volatile; Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Essential oils mouthwash (Active Comparator): 20 ml rinses for 30 seconds with essential oils/2 times daily (1/0/1).
  Interventions: Drug: Essential oils
- essential oils without mouthwash (Experimental): 20 mL rinses for 30 seconds with essential oils without alcohol/2 times daily (1/0/1)
  Interventions: Drug: Essential oils without alcohol
- sterile water mouthwash (Sham Comparator): 20 mL rinses for 30 seconds with sterile water/2 times daily (1/0/1)
  Interventions: Drug: Sterile water

INTERVENTIONS:
Drug: Essential oils
  Other Names: Listerine Mentol
  Arms: Essential oils mouthwash
Drug: Essential oils without alcohol
  Other Names: Listerine Zero
  Arms: essential oils without mouthwash
Drug: Sterile water
  Arms: sterile water mouthwash

SUMMARY:
The accumulation and maturation of oral biofilm in the gingival margin is widely recognised to be the primary aetiological factor in the development of chronic gingivitis. Based on this association, the current treatment of gingivitis is focused on biofilm disruption, which will normally include mechanical processes, both professionally and at home. However, for patients, it is not easy to achieve a proper level of plaque control. The efficient plaque control techniques are very time consuming and require a special motivation and skills for their optimum use. It was at this point where mouthwashes become important, due to the fact that they include diverse types of antimicrobial agents to complement the results of mechanical oral hygiene measures.

The essential oils have been presented as a realiable alternative to the "gold Standard" (Chlorhexidine). However, it use has been limited clinically due to their alcohol contain. Some years ago, a new alternative without alcohol has been launched to the market. This formulation has not been already deeply tested specific antiplaque studies in which the structure of the biofilm remained intact.

The aim of this study was to evaluate the in situ antiplaque effect of 2 antimicrobial agents (based on an essential oils formulation with and without alcohol) in the short term with a posterior analysis on "non-destructured" biofilm with Confocal Laser Scanning Microscope combined with fluorescence staining.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy adults.
* Minimum of 24 permanent teeth.
* No gingivitis (Community Periodontal Index score = 0).
* No periodontitis (Community Periodontal Index score = 0).
* Absence of untreated caries.

Exclusion Criteria:

* Smoker or former smoker.
* Presence of dental prostheses.
* Presence of orthodontic devices
* Antibiotic treatment or routine use of oral antiseptics in the previous 3 months.
* Presence of any systemic disease that could alter the production or composition of saliva.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of bacterial viability | 96 hours after the volunteer has worn the splints with the disks

SECONDARY OUTCOMES:
Thickness in microns | 96 hours after the volunteer has worn the splints with the disks
Percentage of area covered by the biofilm | 96 hours after the volunteer has worn the splints with the disks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quintas V, Prada-Lopez I, Donos N, Suarez-Quintanilla D, Tomas I. Antiplaque effect of essential oils and 0.2% chlorhexidine on an in situ model of oral biofilm growth: a randomised clinical trial. PLoS One. 2015 Feb 17;10(2):e0117177. doi: 10.1371/journal.pone.0117177. eCollection 2015. PMID 25689859